CLINICAL TRIAL: NCT04921839
Title: Awareness of Operating Room Staff About WHO OR Checklist
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Imam Mohammad ibn Saud Islamic University (Other)
Responsible Party: Principal Investigator, mohammad bukhetan alharbi, associate professor, Imam Mohammad ibn Saud Islamic University
Other Study IDs: WHO OR CHECKLIST AWARNESS
Record Dates: First submitted 2021-06-01; First posted 2021-06-10 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Safety Issues
Keywords: WHO checklist; WHO OR ckecklist

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to understand and analyze awareness of proper timing of when to sing in, time out, and sign out for patients who will be operated in Hail multidisciplinary centers, Saudi Arabia. its role in improving communication in OR, and preventing errors. how frequent not comply and potentials of non compliance. how frequent dose WHO OR check list will cause anxiety in the staff, psychological insult ,potentials to be replaced or adjusted according to each specialty needs.

ELIGIBILITY:
Inclusion Criteria: operating room staff of hail region hospitals -

Exclusion Criteria: none

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the survey link will be send to operating room staff through hospital administration, participants bio information is never requested. Informed consent was obtained from all those agreeing to complete a survey. This study was exempt from review board approval at authors' institutions.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
predictive power of respondent on awareness of WHO OR checklist | 20 days
  will include demographics include: gender, specialty, hospital name ,utilization of WHO OR checklist habits, commitment of staff ,communication improvement, its psychological impact over staff, significance potentials, possibility of adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: mohammad alharbi, Study Chair — imam mohamamd ibn saud islamic university
Locations (1):
- Central fourth Health Cluster, Hail, Saudi Arabia